CLINICAL TRIAL: NCT00304733
Title: Wound Healing: Total Contact Cast Vs. Custom-Made Temporary Footwear for Patients With Diabetic Foot Ulceration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rehabilitation Centre Amsterdam (Other)
Collaborators: ConvaTec Inc. (Industry); Ontwikkelingsfonds Orthopedisch maatschoeisel (Unknown)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2024
Record Dates: First submitted 2006-03-16; First posted 2006-03-20 (Estimated); Last update posted 2006-03-20 (Estimated); Status verified 2001-08

CONDITIONS: Neuropathic Foot Ulceration in Individuals With Diabetes
Keywords: neuropathic foot ulcerations - total contact cast - custom -made footwear - off-loading

INTERVENTIONS:
Device: cast vs. shoe

SUMMARY:
Objective: to compare the effectiveness of irremovable total contact casts and custom made temporary footwear to heal neuropathic foot ulcerations in individuals with diabetes

DETAILED DESCRIPTION:
In this prospective clinical trail, 43 patients with plantar ulcer grade 1 or 2 (wagner scale) were randomized to one of two off-loading modalities: total contact cast or custom-made temporary footwear.outcomes assessed were wound surface area reduction (square cm.)and time to wound healing (days0 at 2,4,8 and 16 weeks. to evaluate safety, possible side effects were recorded at each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diabetes
* neuropathic ulcer grade 1/2 (wagner scale)
* confirmed sensory neuropathy

Exclusion Criteria:

* osteomyelitis patients unable to walk
* life threatening co-morbidity ankle/brachial index , 0.4

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43
Dates: Start 2001-08; Study Completion 2005-04

PRIMARY OUTCOMES:
wound surface area reduction

SECONDARY OUTCOMES:
time to wound healing (days)

CONTACTS AND LOCATIONS:
Overall Officials: f. b. van de weg, m.d., Study Chair — rehabiliation centre amsterdam
Locations (1):
- Onze Lieve Vrouwe Gasthuis, Amsterdam, North Holland, Netherlands